CLINICAL TRIAL: NCT03958344
Title: Intraorbital Injection Versus Oral Steroid in Patients With Anterior Idiopathic Orbital Inflammation: A Randomized Clinical Trial
Brief Title: Intraorbital Injection Versus Oral Steroid in Anterior Idiopathic Orbital Inflammation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iran University of Medical Sciences (Other)
Collaborators: Tehran University of Medical Sciences (Other); Mashhad University of Medical Sciences (Other); Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.IUMS.REC.1397.1202
Record Dates: First submitted 2019-05-07; First posted 2019-05-22 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Orbital Pseudotumor
MeSH Terms: conditions — Orbital Pseudotumor | interventions — Prednisolone; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Randomized parallel double arm
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraorbital injection of steroid (Experimental): 2 mL of steroid will be ready for each injection session:
  1 mL Triamcinolone (40 mg) + 1 mL Betamethasone (6 mg) = 2 mL
  For Dacryoadenitis without myositis , 1 mL of this compound will be injected at lacrimal gland through 1 site of injection.
  For Dacryoadenitis plus 1 rectus muscles myositis 1 mL of this compound will be injected at lacrimal gland and 0.5 mL of this compound will be injected at the rectus muscle through 2 separate sites of injection.
  For Dacryoadenitis plus 2 rectus muscles myositis 1 mL of this compound will be injected at lacrimal gland and 0.5 mL of this compound will be injected at either recti muscles through 3 separate sites of injection.
  Interventions: Drug: Triamcinolone + Betamethason
- Oral Steroid (Active Comparator): Each patient will receive oral Prednisolone, 1 mg/kg, for 5-7 days, followed by tapered dose in 12 weeks (according to a pre-defined table of oral administration dose).
  Daily Omeprazole 40mg p.o and daily Calcium Supplement will also be recommended to avoid complications.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Oral Tablet
  Other Names: Oral Prednisolone
  Arms: Oral Steroid
Drug: Triamcinolone + Betamethason — A compound long acting and short acting injectable steroid
  Other Names: Injectable Steroid
  Arms: Intraorbital injection of steroid

SUMMARY:
A multicenter randomised double-arm clinical trial, to compare safety and efficacy of oral versus intralesional injection of steroid in a group of patients suffering from idiopathic orbital inflammation is designed. Outcome measures include number of recurrences, duration of remission, and side effects.

DETAILED DESCRIPTION:
Expected to be finished in 3 years, patient enrollment includes 59 patient in each arm of the study. Inclusion criteria consist of clinical and/or imaging evidence of dacryoadenitis with or without adjacent rectus muscles (superior and inferior recti) myositis. Patients meeting following conditions will be excluded:

1. Age < 15 years
2. Diabetes mellitus
3. Collagen Vascular Diseases
4. Vasculitides
5. Biopsy of lacrimal gland denoting a specific diagnosis (i.e. the term "idiopathic" does not apply)
6. Glaucoma
7. Patients who have lost one eye
8. Bilateral disease
9. Abnormal thyroid-stimulating hormone

Outcome measures include number of recurrences, duration of remission, and side effects.

Patient allocation will be based on blocks of 4. Each patient will undergo lacrimal gland biopsy and subsequently will be allocated to one arm of the study according to a predetermined randomization sequence (balanced block of four). Outcome measures will be recorded in 0, 3 and 6 months after patient enrollment.

Patients in oral steroid group will receive 1 mg/kg/day of Prednisolone, tapered in 3 months (based on a detailed table).

Patients in injection group will receive 1 shot of 1 mL (20 mg Triamcinolone + 3 mg Betamethason) into the lacrimal gland.

ELIGIBILITY:
Inclusion Criteria:

* Dacryoadenitis based on clinical findings and/or imaging with and without adjacent recti muscle myositis

Exclusion Criteria:

* Abnormal thyroid-stimulating hormone
* Systemic Vasculitides
* Bilateral Orbital Inflammation
* Collagen Vascular Diseases
* One Seeing Eye
* Glaucoma
* Diabetes Mellitus

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence number | up to 6 months
  frequency of occurrence of clinical condition showing signs of inflammation recurrence, during or after cessation of steroid therapy
Recurrence time | up to 6 months
  mean time of occurrence of clinical condition showing signs of inflammation recurrence, during or after cessation of steroid therapy
Adverse Effect | up to 6 months
  Any significant ocular or systemic side effect reported by the patient or found in examination sessions

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen B Kashkouli, MD, Principal Investigator — Iran University of Medical Sciences
Locations (1):
- Iran University of Medical Sciences, Tehrān, Tehran Province, Iran

REFERENCES:
- [Background] Swamy BN, McCluskey P, Nemet A, Crouch R, Martin P, Benger R, Ghabriel R, Wakefield D. Idiopathic orbital inflammatory syndrome: clinical features and treatment outcomes. Br J Ophthalmol. 2007 Dec;91(12):1667-70. doi: 10.1136/bjo.2007.124156. Epub 2007 Jul 9. PMID 17620331
- [Background] Bijlsma WR, Paridaens D, Kalmann R. Treatment of severe idiopathic orbital inflammation with intravenous methylprednisolone. Br J Ophthalmol. 2011 Aug;95(8):1068-71. doi: 10.1136/bjo.2010.195552. Epub 2011 Feb 24. PMID 21349945
- [Result] El Nasser A Mohammad A. Local steroid injection for management of different types of acute idiopathic orbital inflammation: an 8-year study. Ophthalmic Plast Reconstr Surg. 2013 Jul-Aug;29(4):286-9. doi: 10.1097/IOP.0b013e318293750c. PMID 23839634
- [Result] Leibovitch I, Prabhakaran VC, Davis G, Selva D. Intraorbital injection of triamcinolone acetonide in patients with idiopathic orbital inflammation. Arch Ophthalmol. 2007 Dec;125(12):1647-51. doi: 10.1001/archopht.125.12.1647. PMID 18071116
- [Result] Reggie S, Neimkin M, Holds J. Intralesional corticosteroid injections as treatment for non-infectious orbital inflammation. Orbit. 2018 Feb;37(1):41-47. doi: 10.1080/01676830.2017.1353110. Epub 2017 Sep 5. PMID 28872378